CLINICAL TRIAL: NCT04938336
Title: Evaluation of a Decision Aid Tool in Rectal Cancer patiënts
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Sint-Lucas Gent (Other); AZ Sint-Jan AV (Other); AZ Delta (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10030
Record Dates: First submitted 2021-06-01; First posted 2021-06-24 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
Keywords: low anterior resection syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- expert healthcare professionals: Delphi Procedure
  Interventions: Behavioral: Delphi Procedure and interviews
- healthcare professionals, patients and informal carers: interviews
  Interventions: Behavioral: Delphi Procedure and interviews

INTERVENTIONS:
Behavioral: Delphi Procedure and interviews — Delphi procedure with expert healthcare professionals and interviews with patients, healthcare professionals and informal carers

SUMMARY:
Adapt and evaluate a decision aid for patients with rectal cancer. Phase 1 : decision aid testing (Delphi) multicentric Phase 2: pilot test decision aid

DETAILED DESCRIPTION:
Adapt and evaluate a decision aid for patients with rectal cancer. Phase1: decision aid testing (Delphi) A pilot version of the Belgian decision aid was developed and validated through a double Delphi procedure. In this study, the assessment is extended to several multicentre experts. The panel consists of ten experts who have extensive knowledge in the field of rectal cancer or scientific research. They are asked to evaluate the information and questions on accuracy, clarity, readability and relevance. They score the items of the decision aid using a 4-point Likert-type scale (one (one = totally irrelevant; four = very relevant) and a dichotomous scale (one = clear, two = not clear) to assess relevance and clarity of wording, respectively (see Appendix 2 to this application). To quantify the degree of content validity, the Content Validity Index (CVI) is used.

Phase2: pilot test decision aid The final step of the study is a pilot test of the decision aid with patients who will undergo surgery/watch and wait strategy in the near future and with healthcare professionals who work with the decision aid. The aim is to test the acceptability of the decision aid with the patient and the ease of use with the healthcare professional. With the feedback from the patients and the healthcare professional, the decision aid can be further refined.

During the consultation in which the intervention is discussed, the consent to participate will be asked of the patient and also of the informal carer who may be present at that moment. Participation in the study means that during this consultation, the caregiver involved will go through the decision aid completely with the patient and any informal carer. After the intervention, they will be asked to give feedback on their experiences with the use of the decision aid. This will be done by means of an interview for the patients, informal carers and care workers involved. The interview with the patient (and informal carer if applicable) will take place at home or in the hospital, depending on their preference. The interview with the caregiver takes place in the hospital where the caregiver works. If the current Covid-19 pandemic does not allow for a visit to the patient's home or to another hospital, the interviews will be conducted by telephone or video call.

ELIGIBILITY:
Delphi procedure

Inclusion Criteria:

* expert healthcare professionals caring for patients with rectal cancer

Exclusion Criteria:

* none

Interviews Inclusion criteria

* Patients in which the decision aid was tested
* patients with a tumor in the last 10cm of the rectum
* healthcare professionals who have used the decision aid tool
* informal carer indicated by the patient Exclusion
* patients who have no treatment choice due to oncological reasons

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with rectal cancer healthcare professionals caring for patients with rectal cancer informal carers of patients with rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Assessment of accuracy of the decision aid tool trough a delphi procedure | 2-3 months (until consensus)
  Assessment of accuracy of the decision aid tool through a delphi procedure
Assessment of clarity of the decision aid tool trough a delphi procedure | 2-3 months (until consensus)
  Assessment of clarity of the decision aid tool trough a delphi procedure
Assessment of relevance of the decision aid tool trough a delphi procedure | 2-3 months (until consensus)
  Assessment of relevance of the decision aid tool trough a delphi procedure
Assessment of readability of the decision aid tool trough a delphi procedure | 2-3 months (until consensus)
  Assessment of readability of the decision aid tool trough a delphi procedure
Assessment of the acceptability of the decision aid tool through individual interview | about 60 minutes
  Assessment of the acceptability of the decision aid tool through individual interview
Assessment of the usability of the decision aid tool through individual interviews | about 60 minutes
  Assessment of the usability of the decision aid tool through individual interviews

CONTACTS AND LOCATIONS:
Overall Officials: Piet Pattyn, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University hospital Ghent, Ghent, Oost-Vlaanderen
  - University Hospital Ghent, Ghent